CLINICAL TRIAL: NCT05999305
Title: The Effects of Using an Escape Room Game to Improve Senior Nursing Students' Critical Thinking Dispositions and Skills in Vietnam
Brief Title: Using an Escape Room Game in Teaching the Critical Care Nursing Course
Acronym: ER_Game
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: N202307017
Record Dates: First submitted 2023-08-13; First posted 2023-08-21 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-08

CONDITIONS: Critical Thinking
Keywords: thinking; escape; nursing; student

STUDY DESIGN:
Intervention Model Description: Two teaching methods in the Critical Care Nursing course will be implemented including the conventional teaching combining an escape room game and the conventional class with case-based teaching.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The intervention group (Experimental): The conventional class and an escape room game will be implemented for the intervention.
  Interventions: Other: Teaching the critical care nursing course with an Escape Room game
- The comparison group (Active Comparator): The conventional class and a case-based learning will be implemented for the comparison
  Interventions: Other: Teaching the critical care nursing course with a case-based learning

INTERVENTIONS:
Other: Teaching the critical care nursing course with an Escape Room game — A teacher will begin with a 1.5-hour lecture, followed by an escape room game to reinforce learning through case studies for another 1.5 hours. The first section of the game will be a ten-minute pre-brief. The game will then begin promptly at a designated time and will be played in groups of six to seven students, with each group seated separately in a classroom. The game will last up to fifty minutes, during which all groups will be assisted to complete puzzles within the time limit. After the game, a fifteen-minute debriefing session will be held by the teacher, during which the students will reflect on their performance and what they learned about the cases and related topics. The teacher will finally provide feedback and support to the groups during this session.
  Arms: The intervention group
Other: Teaching the critical care nursing course with a case-based learning — Students in the comparison group will also receive a 1.5 hour lecture which is the same as those in the intervention group. Another 1.5 hour is a case-based learning session, with six sessions in total over six weeks. The case-based learning sessions will include a pre-brief, teamwork, and debrief, and will be facilitated by the same teacher and teaching assistant and will primarily be provided with paper-based case studies.
  Arms: The comparison group

SUMMARY:
Critical thinking is one of the most desired outcomes of nursing education worldwide. The impact of game-based learning, including the use of an escape room game, on the development of critical thinking ability in nursing students remains uncertain. The main purpose of this study is going to evaluate an escape room game as a learning method in Critical Care Nursing course in improving senior nursing students' critical thinking dispositions and skills. In addition to the main purpose, this study also aims to investigate the effects of incorporating an escape room game into a Critical Care Nursing course in improving senior nursing students' knowledge about critical care nursing, learning motivation, and satisfaction with the learning method. This is a two-arm parallel randomized controlled trial conducted on senior nursing students at Tra Vinh University in Vietnam. Two teaching methods in the Critical Care Nursing course will be applied.

DETAILED DESCRIPTION:
Critical thinking is one of the most desired outcomes of nursing education worldwide. The impact of game-based learning, including the use of an escape room game, on the development of critical thinking ability in nursing students remains uncertain.

The main purpose of this study is going to evaluate an escape room game as learning method in Critical Care Nursing course in improving senior nursing students' critical thinking dispositions and skills. In addition to the main purpose, this study also aims to investigate the effects of incorporating an escape room game into a Critical Care Nursing course in improving senior nursing students' knowledge about critical care nursing, learning motivation, and satisfaction with the learning method.

This a two-arm parallel randomized controlled trial conducted on senior nursing students at Tra Vinh University in Vietnam. Two teaching methods in the Critical Care Nursing course will be applied. A conventional class with an escape room game will be implemented for the intervention group while a conventional class with case-based learning will be the teaching method for the comparison group.

The study will be a repeated-measurement design with three time points. Mean, standard deviation, frequency, percentage, t-test, and chi-squared test will be conducted. Generalized Estimating Equations will be used to analyze the intervention effect and time effect on scores of critical thinking dispositions and skills, knowledge of critical care nursing, and learning motivation over three-time points. Generalized Estimating Equations will also allow us to explore the interaction between group and time, as well as control for any potential covariates. The intention of this study is that its findings will offer valuable insights for faculty members to consider incorporating escape room games into their teaching methodologies.

ELIGIBILITY:
Inclusion Criteria:

* Nursing students who are in their senior year in the bachelor program and take Critical Care Nursing which is a required course.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2023-09-08 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
The critical thinking skills of nursing students | The measurement will be repeated in three time points including the pre-test, immediately after the completion of the teaching course, and one month after the completion of the teaching course
  The Critical Thinking Self-Assessment Scale (CTSAS) will be used to assess the critical thinking skills of nursing students. This 46-item scale is scored on a six-point Likert scale of 0 to 6, with 0 corresponding to "never" and 6 to "always." The total scores range from 0 to 276, with a higher score indicating a higher level in critical thinking skills.
The critical thinking disposition of nursing students | The measurement will be repeated in three time points including the pre-test, immediately after the completion of the teaching course, and one month after the completion of the teaching course
  The Critical Thinking Disposition Scale (CTDS) will measure the critical thinking disposition of nursing students. The CTDS has 11 items with five-point Likert-type responses (1 = strongly disagree; 5 = strongly agree). The total scores range 11-55 for the scale, with 7-35 for the critical openness scale (the first seven items) and 4-20 for reflective skepticism (the last four items). The higher score indicates a better disposition of critical thinking.

SECONDARY OUTCOMES:
The knowledge about Critical Care Nursing of nursing students | The measurement will be repeated in three time points including the pre-test, immediately after the completion of the teaching course, and one month after the completion of the teaching course
  The retention of students' knowledge about Critical Care Nursing will be evaluated through a structured questionnaire. It will consist of thirty multiple-choice questions, covering six topics of the course. Participants will select one answer or "don't know" per question. Each correct response will be scored one points and incorrect response or "don't know" will be scores zero points, resulting in a total score
Student's learning motivation | The measurement will be repeated in three time points including the pre-test, immediately after the completion of the teaching course, and one month after the completion of the teaching course
  The Motivated Strategies for Learning Questionnaire (MSLQ) will be used to assess the students' learning motivation. This 31-item instrument is a 7-point Likert scale, ranging from 1 (not at all true of me) to 7 (very true of me). The total scores range from 31 to 217 with a higher score indicating a higher motivation level.
Students' satisfaction with the course. | The measurement will be conducted immediately after the completion of the teaching course.
  The 13-item student satisfaction questionnaire was developed to assess students' satisfaction with the teaching method and also their experience with the learning activities throughout the course. This is a 5-point Likert scale (ranging from 1 = strongly disagree to 5 = strongly agree). The total score ranges from 13 to 65, with higher scores indicating a higher level of satisfaction.
The Escape Room Perception of nursing students | The measurement will be conducted immediately after the completion of the teaching course.
  The Escape Room Perception Scale (ERPS) will be used to evaluate the perception of nursing students about the escape room game, including its effectiveness in supporting their learning, the nature of the learning activity, and the team learning. The perception scale includes twelve items and is a five-point Likert scale ranging from "1 = strongly disagree" to "5 = strongly agree." The higher scores that participants achieve, the more satisfied they will feel about a game, and also indicating the effectiveness of the escape room game.

CONTACTS AND LOCATIONS:
Overall Officials: Yeu-Hui Chuang, Professor, Principal Investigator — School of Nursing, College of Nursing of Taipei Medical University
Locations (1):
- Nursing Department of Tra Vinh University, Thành phố Trà Vinh, Vietnam

IPD SHARING:
Plan to Share IPD: No
The detailed description of this study and outcomes as well